CLINICAL TRIAL: NCT02099266
Title: A Pilot Study to Determine the Safety and Efficacy of Using Hyperbaric Oxygen Therapy to Improve Umbilical Cord Blood Stem Cell Homing and Subsequent Engraftment
Brief Title: Use of Hyperbaric Oxygen Therapy to Improve Umbilical Cord Blood Stem Cell Homing and Subsequent Engraftment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT-2011-08-01
Record Dates: First submitted 2014-03-20; First posted 2014-03-28 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome (MDS); Hodgkins Lymphoma; Non-Hodgkins Lymphoma
Keywords: Umbilical Cord Blood (UCB) Stem Cell Transplant; Hyperbaric oxygen; Leukemia; Lymphoma; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hyperbaric Oxygen Treatment (Experimental): Administration of hyperbaric oxygen the morning of UCB transplant.
  Interventions: Device: Administration of hyperbaric oxygen

INTERVENTIONS:
Device: Administration of hyperbaric oxygen — Hyperbaric oxygen at 2.5 atmospheres absolute (ATA) for a total of 2 hours
  Other Names: Monoplace Hyperbaric Chamber Model 3200 and 3200R

SUMMARY:
By doing this study, researchers hope to learn the following:

* If providing hyperbaric oxygen (HBO) therapy prior to an umbilical cord blood (UBC) transplant will help to improve the homing process
* The safety of HBO administration in the setting of the UBC transplant
* The effects of HBO therapy on the engraftment process

DETAILED DESCRIPTION:
Research has suggested that high levels of erythropoietin (EPO) decreases the ability of infused umbilical cord stem cells to home to the bone marrow. The investigators will investigate the use of hyperbaric oxygen (HBO) therapy to decrease the plasma concentrations of EPO prior to UBC transplant and evaluate the resulting impact on UBC homing.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Subjects must be >/= 17 yrs and </= 70 yrs for non-myeloablative transplant
* Subjects must be >/= 17 yrs and </= 55 yrs for myeloablative transplant
* Subjects with Acute Myeloid Leukemia (AML), Acute Lymphoblastic Leukemia (ALL), Myelodysplastic Syndrome (MDS), Hodgkin's Lymphoma (HL) and Non-Hodgkin's Lymphoma (NHL) who are considered for UCB transplant
* Use of approved form of contraception
* Karnofsky performance status of >/= 70%
* Adequate hepatic, renal, pulmonary and cardiac function. Criteria include:
* ALT (alanine aminotransferase), AST (aspartate aminotransferase: < 4x IULN (institutional upper limit of normal)
* Total bilirubin </= 2 mg/dL
* Serum creatinine < 2.0 mg/dL
* Left ventricular ejection fraction >/= 45%
* FEV1 (forced expiratory volume), FVC (forced vital capacity) and DLCD (diffusing capacity of lung for carbon monoxide) >/= 50% of predicted value (corrected to serum hemoglobin)

Exclusion Criteria:

* Pregnancy or breast feeding
* Severe chronic obstructive pulmonary disease requiring oxygen supplementation
* History of spontaneous pneumothorax
* History of seizures
* Claustrophobia
* Asthma
* Uncontrolled viral or bacterial infection at the time of enrollment
* Active or recent (prior 6 months) invasive fungal infection without interdisciplinary consult and approval

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Aljitawi OS, Paul S, Ganguly A, Lin TL, Ganguly S, Vielhauer G, Capitano ML, Cantilena A, Lipe B, Mahnken JD, Wise A, Berry A, Singh AK, Shune L, Lominska C, Abhyankar S, Allin D, Laughlin M, McGuirk JP, Broxmeyer HE. Erythropoietin modulation is associated with improved homing and engraftment after umbilical cord blood transplantation. Blood. 2016 Dec 22;128(25):3000-3010. doi: 10.1182/blood-2016-05-715292. Epub 2016 Oct 19. PMID 27760758

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperbaric Oxygen Treatment
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hyperbaric Oxygen Treatment
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 13
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety of HBO Administration in the Setting of UCB Stem Cell Transplantation
Description: Treatment limiting toxicities are defined as the occurrence of any of the following complications within 24hrs of treatment: pneumothorax, death, irreversible grade III or any grade IV toxicity that is determined by the treating physician to be related to HBO therapy.
Time Frame: Toxicity assessment with 24hrs of treatment
Population: One patient treatment was shortened by approximately 10 minutes because of nausea attributed to concomitant medications.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Treatment
Number analyzed (Participants) | 15
Participants
  grade IV leukopenia | 15
  grade III/IV neutropenia | 12
  grade III/IV anemia | 12
  grade III/IV thrombocytopenia | 13

2. Secondary Outcome: Determine the Effects of HBO Therapy on Neutrophil Count Recovery.
Description: Time in days until neutrophil count recovery is achieved; neutrophil count recovery is defined as three consecutive days of achieving a neutrophil level >/= 500 u/L.
Time Frame: Daily measurement of neutrophil counts up to 90 days post transplant.
Measure: Median (Full Range); unit: Days
Groups:
- Reduced-Intensity Conditioning: Reduced-Intensity (also referred to as: "Non-myeloablative") transplant patients will receive the following chemotherapeutic agents and radiation on the respective days:
  Day -6 : fludarabine 40mg/m2 (milligram per meter squared) intravenously (IV), cyclophosphamide 50mg/kg IV, and mesna 50mg/kg IV Day-5 to -2: fludarabine 40mg/m2 intravenously (IV) Day -1: Total body irradiation (TBI) 200 centrigray (cGy)
- Myeloablative Conditioning: Myeloablative transplant patients will receive the following chemotherapeutic agents and radiation on the respective days:
  Day -10, -9, and -8: Fludarabine (25 mg/m2 IV) IV Day -7, -6, -5, and -4: Total body irradiation 165 cGy twice daily Day -3 and -2: Cyclophosphamide (60 mg/kg/day ) and mesna 50mg/kg/day (milligrams per kilogram per day) IV
Arm/Group | Reduced-Intensity Conditioning | Myeloablative Conditioning
Number analyzed (Participants) | 9 | 6
Days | 7 [6 to 17] | 24.5 [16 to 45]

3. Secondary Outcome: Proportion of Reduced Intensity Conditioning Participants With Complete Engraftment.
Description: Complete engraftment is defined as as marrow reconstitution of greater than 90% of donor cells. Degree of engraftment will be determined through bone marrow chimerism assessment at either day 21 or day 28.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Conditioning
Number analyzed (Participants) | 9
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse clinical events experienced by participants will be collected and reported from initiation of HBO treatment and through engraftment or day +90, whichever comes first.
Arm/Group | Hyperbaric Oxygen Treatment
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperbaric Oxygen Treatment (N=15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Respiratory infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperbaric Oxygen Treatment (N=15)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2)
Anal pain (Gastrointestinal disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 12 (87)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 (5)
Blood bilirubin increased (Investigations) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (3)
Chills (General disorders) | 6 (6)
Concentration impairment (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (13)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Edema face (General disorders) | 2 (3)
Edema limbs (General disorders) | 6 (10)
Edema trunk (General disorders) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 2 (6)
Eye pain (Eye disorders) | 1 (2)
Facial pain (General disorders) | 2 (2)
Fatigue (General disorders) | 8 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (7)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 2 (3)
Flushing (Vascular disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 6 (9)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 7 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (11)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 6 (9)
Infusion related reaction (General disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Malaise (General disorders) | 5 (5)
Menorrhagia (Reproductive system and breast disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (16)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 12 (70)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 4 (4)
Pain (General disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
platelet count decreased (Investigations) | 14 (114)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (12)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 (3)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (1)
Scleral disorder (Eye disorders) | 2 (2)
Sepsis (Renal and urinary disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Infections and infestations) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (6)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (3)
Tremor (Nervous system disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 (4)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 15 (86)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes